CLINICAL TRIAL: NCT03755856
Title: A Survivorship Project to UnerstAnd and to impRove Long-Term Outcomes for Acute Myeloid Leukemia Patients (SPARTA): the Sparta Platform
Brief Title: Long-term Outcomes for Acute Myeloid Leukemia Patients
Acronym: 1621-QLG-LG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: GIMEMA-EORTC 1621-QLG-LG
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Health-related quality of life

SUMMARY:
This international observational study aims at examining the patterns of health-related quality of life differences between long-term acute myeloid leukemia patients and their healthy peers from the general population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of all subtypes of de novo AML, according to WHO criteria (at least 20% blasts in the bone marrow), except acute promyelocytic leukemia (APL).
* Age at AML diagnosis ≥ 18 years,
* Date of AML diagnosis at least 5 years before study enrollment,
* AML-free status at study enrollment,
* Written informed consent provided.

Exclusion Criteria:

* Major cognitive deficit or psychiatric problems hampering a self-reported evaluation,
* Not speaking and reading the language of the participating country,
* More than 75 years at the time of study enrollment,
* Receiving any active treatment for AML at the time of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study patients are acute myeloid leukemia long-term survivors
Sampling Method: Non-Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of differences in SF-36 scores | At enrollment
  The Role Physical scores of AML survivors will be compared to that in the general population as assessed by SF-36 questionnaire. Comparisons will be performed on age-sex matched pairs of AML patients and healthy subjects from the general population.

SECONDARY OUTCOMES:
Outcomes from SF-36 questionnaire will be described and compared between AML patients from RCTs vs non RCTs. | At enrollment
  Prior to these comparisons, to further minimize the possible influence of confounding factors, RCTs and non RCTs AML groups will be previously matched on their estimated propensity scores
QoL profiles of AML survivors will be compared with those in the general population also as assessed by EORTC QLQ-C30 questionnaire. | At enrollment
  Comparisons will be adjusted by age and sex, using the European reference values for the EORTC QLQ-C30. A subgroup analysis on elderly patients (i.e. 60+ patients) will be also performed.
Outcomes from SCQ questionnaire will be described and compared between AML patients from RCTs vs non RCTs. | At enrollment
  Prior to these comparisons, to further minimize the possible influence of confounding factors, RCTs and non RCTs AML groups will be previously matched on their estimated propensity scores.
Outcomes from EORTC QLQ-C30 questionnaire will be described and compared between AML patients from RCTs vs non RCTs. | At enrollment
  Prior to these comparisons, to further minimize the possible influence of confounding factors, RCTs and non RCTs AML groups will be previously matched on their estimated propensity scores.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, Study Chair — GIMEMA Foundation; Frédéric Baron, Study Director — European Organisation for Research and Treatment of Cancer - EORTC
Locations (39):
- Belgium (3):
  - UZ Gasthuisberg, Leuven
  - CHR Citadelle-CHU, Liège
  - University of Liège, Liège
- Croatia (2):
  - KBC Rijeka, Rijeka
  - University Hospital Centre Zagreb, Zagreb
- Les Hôpitaux Universitaires de Strasbourg, Lyon, France
- Italy (29):
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. LANCISI - G. SALESI, Ancona
  - U.O. Ematologia con trapianto - Azienda Ospedaliero-Universitaria Policlinico di Bari, Bari
  - UOC Ematologia Ospedale " Monsignor Raffaele Dimiccoli", Barletta
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Divisione clinicizzata di Ematologia - Dipartimento di Scienze Mediche - Osp. Ferrarotto, Catania
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Cona
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - IRCCS_AOU San Martino-IST.Clinica Ematologica, Genova
  - Milano Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - UOC di Ematologia-Centro Emofilia e Trombosi - Ospedale Ascalesi - ASL Napoli 1, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Orbassano Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - U.O. di Ematologia con trapianto - A.U. Policlinico "Paolo Giaccone", Palermo
  - U.O. Ematologia e CTMO- AOU di Parma, Parma
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Ematologia - Ospedale San Carlo, Potenza
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Divisione di Ematologia - Ospedale S.Eugenio, Roma
  - Ematologia Policlinico - Università degli Studi di Roma Tor Vergata (PTV), Roma
  - Istituto di Semeiotica Medica - Ematologia - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Roma Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Università degli Studi "Sapienza" - Dip Medicina di Precisione e Ricerca Traslazionale UOC Ematologia, Roma
  - U.O. di Ematologia - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ematologia - AOU Sassari, Sassari
  - Torino Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
- University Clinic of Hematology-Skopje, Skopje, North Macedonia
- University hospital Bratislava, Bratislava, Slovakia
- UKC Ljubljana, Ljubljana, Slovenia
- Ankara University School Of Medicine Cebeci Campus Adult Hematology Department and BMT Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided